CLINICAL TRIAL: NCT06691906
Title: A Clinical Study to Evaluate the Relative Bioavailability of MK-0616 Formulations in Healthy Adult Participants
Brief Title: A Clinical Study of Enlicitide Decanoate (MK-0616) in Healthy Adult Participants (MK-0616-025)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 0616-025; MK-0616-025 (Other: MSD)
Record Dates: First submitted 2024-11-13; First posted 2024-11-18 (Actual); Last update posted 2024-11-18 (Actual); Status verified 2024-11

CONDITIONS: Healthy
MeSH Terms: interventions — MK-0616

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Enlicitide Decanoate Treatment A (Experimental): Participants will receive a single dose of enlicitide decanoate formulation 1 on Day 1 on an empty stomach.
  Interventions: Drug: Enlicitide decanoate
- Enlicitide Decanoate Treatment B (Experimental): Participants will receive a single dose of enlicitide decanoate formulation 2 on Day 1 on an empty stomach.
  Interventions: Drug: Enlicitide decanoate

INTERVENTIONS:
Drug: Enlicitide decanoate — Oral tablet
  Other Names: MK-0616

SUMMARY:
The purpose of this study is to learn what happens to the amount of enlicitide decanoate in the blood when enlicitide decanoate is given in different formulations.

ELIGIBILITY:
Inclusion Criteria:

* Continuous non-smoker who has not used nicotine- and tobacco-containing products for at least 3 months prior to the first dosing.
* Medically healthy with no clinically significant medical history.

Exclusion Criteria:

* Has a history of gastrointestinal disease or has had a gastric bypass or similar surgery.
* Has a history of cancer (malignancy).

Ages: 19 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2024-03-18 (Actual); Primary Completion 2024-05-01 (Actual); Study Completion 2024-05-01 (Actual)

PRIMARY OUTCOMES:
Area Under the Concentration-Time Curve from 0 to 24 hours (AUC0-24) of enlicitide decanoate | Predose and at designated timepoints (up to 24 hours postdose)
  Blood samples will be collected to determine the AUC0-24 of enlicitide decanoate.
Area Under the Concentration-Time Curve from 0 to Time of Last Quantifiable Sample (AUC0-last) of enlicitide decanoate | Predose and at designated timepoints (up to 168 hours postdose)
  Blood samples will be collected to determine the AUC0-last of enlicitide decanoate.
Area Under the Concentration-Time Curve from 0 to Infinity (AUC0-inf) of enlicitide decanoate | Predose and at designated timepoints (up to 168 hours postdose)
  Blood samples will be collected to determine the AUC0-inf of enlicitide decanoate.
Maximum Plasma Concentration (Cmax) of enlicitide decanoate | Predose and at designated timepoints (up to 168 hours postdose)
  Blood samples will be collected to determine the Cmax of enlicitide decanoate.
Time to Maximum Plasma Concentration (Tmax) of enlicitide decanoate | Predose and at designated timepoints (up to 168 hours postdose)
  Blood samples will be collected to determine the Tmax of enlicitide decanoate.
Apparent Terminal Half-Life (t1/2) of enlicitide decanoate | Predose and at designated timepoints (up to 168 hours postdose)
  Blood samples will be collected to determine the t1/2 of enlicitide decanoate.
Apparent Clearance (CL/F) of enlicitide decanoate | Predose and at designated timepoints (up to 168 hours postdose)
  Blood samples will be collected to determine the CL/F of enlicitide decanoate.
Apparent Volume of Distribution During Terminal Phase (Vz/F) of enlicitide decanoate | Predose and at designated timepoints (up to 168 hours postdose)
  Blood samples will be collected to determine the Vz/F of enlicitide decanoate.

SECONDARY OUTCOMES:
Number of Participants Who Experience an Adverse Event (AE) | Up to approximately 44 days
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of the study intervention, whether or not considered related to the study intervention.
Number of Participants Who Discontinue Study Treatment Due to an AE | Up to approximately 44 days
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of the study intervention, whether or not considered related to the study intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (1):
- Celerion (Site 0001), Lincoln, Nebraska, United States

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- See also: Merck Clinical Trials Information — http://www.merckclinicaltrials.com